CLINICAL TRIAL: NCT05392686
Title: Single Arm, Single Center, Phase II Clinical Study of First-line in PD1 and PARP for Maintenance Therapy for Advanced Non-small Cell Lung Cancer (Lung Squamous Cell Carcinoma)
Brief Title: PD1 and PARP for Maintenance Therapy in NSLLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20220325
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
Keywords: pd1; PARP
MeSH Terms: conditions — Lung Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Immune Checkpoint Inhibitors; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: PD1 + PARP (Experimental): For the Induction Phase, participants receive 4 cycles:
  PD1 200 mg, intravenous (IV) on Day 1 of each 21-day cycle PLUS carboplatin PLUS a taxane (either paclitaxel or nab-paclitaxel) for 4 cycles (21-day cycles). If the participant has a complete or partial response or stable disease to induction therapy, the participant to maintenance therapy.
  For the Maintenance Phase, participants receive PD1 IV on Day 1 of each 21-day for up to 31 cycles PLUS maintenance oral PARP 100 mg twice daily. Until centrally verified progressive disease, physician decision or intolerable toxicity.
  Interventions: Drug: PD-1 inhibitor; Drug: PARP inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — Tirelizumab
Drug: PARP inhibitor — Fluzopari capsule

SUMMARY:
PARP inhibitor and PD1 in lung squamous cell carcinoma The current study will compare PD1 plus maintenance PARP for the treatment of squamous NSCLC. The study's 2 primary hypotheses are: respect to progression-free survival (PFS) per RECIST 1.1 by blinded independent clinical review (BICR).

Overall survival (OS).

DETAILED DESCRIPTION:
This study has 2 phases: an Induction Phase (4 Cycles) and a Maintenance Phase (Up to 31 cycles ). In the Induction Phase, participants receive pd1 plus carboplatin plus a taxane (paclitaxel or nab-paclitaxel). In the Maintenance Phase, participants with a partial or complete disease response or with stable disease after completing four cycles of induction therapy and who meet eligibility criteria will be randomly assigned to receive PD1 plus maintenance PAPR. In the Maintenance Phase, participants randomly assigned to receive pembrolizumab for up to 31 cycles plus maintenance until centrally verified progressive disease (PD), intolerable toxicities, or physician decision."

ELIGIBILITY:
Inclusion Criteria:

* 1 NSCLC confirmed by pathology (histology or cytology)

  2. First line treatment of patients with immune combined with chemotherapy into immune maintenance treatment;

  3. 18-75 years old, both male and female;

  2. There are stage IIIA, IIIB or IIIc NSCLC diagnosed according to the 8th edition of the American Joint Committee on cancer.

  3. Stage III NSCLC that cannot undergo radical surgery was confirmed and recorded by the multidisciplinary tumor committee or the treating physician in consultation with the thoracic surgeon.

  4. In the whole body fluorodeoxyglucose (FDG) - pet or FDG-PET / CT and diagnostic quality CT or MRI scans of the chest, abdomen, pelvis and brain, there was no evidence of metastatic disease as stage IV NSCLC.

Note: unless otherwise demonstrated, the presence of pleural / pericardial effusion is considered to indicate metastatic disease. For pleural effusion in both CT chest scan and frontal chest X-ray examination, pleural puncture is required to confirm that the pleural effusion is cytologically negative. Participants whose effusion was exudate were excluded, even if their effusion was cytologically negative. Subjects who have met the remaining inclusion / exclusion criteria, and pleural effusion is not visible on chest X-ray examination in front and side views, or there is too little effusion to be safely extracted can enter the study.

5. Having a measurable disease as defined in RECIST 1.1, at least one lesion is suitable as a target lesion (determined by the investigator / imaging review of the local research center).

4. No more than 28 days before the first study, CT or MRI scan, at least one previous target lesion without radiotherapy (recistv1.1).

5. No previous treatment (chemotherapy, targeted therapy or radiotherapy) for stage III NSCLC.

6. ECoG physical fitness status is 0 or 2 points.

7. Life expectancy is at least 12 weeks.

8. No antiangiogenic drugs or PARP inhibitors have been used in previous treatment;

9. All acute toxic reactions caused by previous anti-tumor treatment or surgery are relieved before the screening period

Level 10.0-1 (judged according to NCI CTCAE 5.0) or to the level specified in the inclusion / exclusion criteria

(except for hair loss and other toxicity that the researchers believe does not pose a safety risk to the subject).

11. No blood transfusion and blood products were used within 14 days before the first administration, and G-CSF and other hematopoietic stimulating factors were not used for correction.

12. Before the first drug study, the laboratory test values meet the following conditions:

1. Blood routine:

   White blood cell count (WBC) ≥ 3.0 × 109/L；

   Absolute neutrophil count (ANC) ≥ 1.5 × 109/L；

   Platelet (PLT) ≥ 100 × 109/L；

   Hemoglobin content (Hgb) ≥ 9.0 g / dl;
2. Liver function:

   Aspartate aminotransferase (AST) ≤ 2.5xuln in subjects without liver metastasis,

   Alanine liver aminotransferase (ALT) ≤ 2.5x ULN;

   ALT and AST of patients with liver metastasis were < 5xuln;

   Serum total bilirubin (TBIL) ≤ 1.5xuln (excluding Gilbert syndrome, total bilirubin < 3.0mg/dl); Albumin (ALB) ≥ 3G / dl;
3. Renal function:

   Serum creatinine ≤ 1.5xuln or creatinine clearance rate (CrCl) ≥ 40ml / minute
4. Coagulation function:

   International standardization ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
5. Others:

   Lipase ≤ 1.5xuln. If lipase > 1.5xuln but there is no clinical or imaging confirmed pancreatitis, it can be included in the group;

   Amylase ≤ 1.5xuln. If amylase > 1.5xuln but there is no clinical or imaging confirmed pancreatitis, it can be included in the group.

   Alkaline phosphatase (ALP) ≤ 2.5uln, ALP ≤ 5uln in subjects with bone metastasis;

   13. For female subjects of childbearing age who are not sterilized surgically, the serum hCG test must be negative and non lactating within 3 days before the first medication. Contraceptive drugs must be used by male subjects within 6 months after the end of the reproductive age;

   14. The subjects voluntarily joined the study, with good compliance, safety and survival follow-up.

   Exclusion Criteria:
   1. Suffering from small cell lung cancer or mixed tumor with small cell components. Note: subjects with squamous NSCLC are not eligible for pemetrexed containing chemotherapy.
   2. Have a history of MDS / AML, current diagnosis or characteristics suggestive of these diseases.
   3. Weight loss > 10% (from baseline) has been recorded in the past 3 months.
   4. There is a radiotherapy plan, in which the volume (V20) of the whole lung (whole lung v20-gtv) with a total radiation dose of > 20 Gy may exceed that of the lung. 34% of the volume. Note: subjects must be evaluated by a radiation oncologist during screening.
   5. received previous chest radiotherapy, including radiotherapy for esophageal, mediastinal or breast cancer.
   6. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs targeting another stimulatory or co inhibitory T cell receptor (e.g. CTLA-4, OX-40, CD137).
   7. Previous treatment with fluzopari or any other PARP inhibitor.
   8. Major surgery (other than vascular access implantation) was performed within 4 weeks before the first administration of the study drug. Note: if the subject has had major surgery or vascular access implantation, he must have fully recovered from therapeutic toxicity and / or complications before starting the study intervention.
   9. It is expected that any other form of antitumor treatment will be required during the study period.
   10. Have received live vaccine within 30 days before the first administration of the test drug. Examples of live vaccines include, but are not limited to, the following vaccines: measles, mumps, rubella, chickenpox / shingles (varicella), yellow fever, BCG and typhoid vaccines. Since seasonal influenza vaccines for injection are usually inactivated virus vaccines, they are allowed to be used; But intranasal influenza vaccines (e.g., FluMist ®） It is a live attenuated vaccine, so it is not allowed to be used.

   11Strong inducers of CYP3A4 (phenobarbital, enzalutamide, phenytoin, rifampicin, rifampicin, rifapentine, carbamazepine, nevirapine and St. John's grass) or medium inducers (e.g. bosentan, faviren and modafinil) that cannot be stopped during the study period are currently being received. Before starting fluzopari treatment, pentobarbital needs a 5-week washout period, and other drugs need a 3-week washout period.

   12At present, they are receiving potent inhibitors of cytochrome P450 (CYP) 3A4 (such as itraconazole, telithromycin, clarithromycin, protease inhibitors strengthened with ritonavir or kirostat, indinavir, saquinavir, nefinavir, bosepovir, terapivir) or intermediate inhibitors (such as ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) that cannot be stopped during the study period. The elution period required before starting fluzopari is 2 weeks.

   13 The dose of piroxicam (e.g. at least 2.5 days before or after administration of piroxicam) and other drugs other than piroxicam (at least 2.5 days after administration of NSD).

   14 In the judgment of the investigator, resting electrocardiogram (ECG) indicates uncontrolled and potentially reversible heart disease (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, electrolyte disorder, etc.), or the subject has congenital long QT syndrome.

   15 Having a diagnosis of immune deficiency or being treated with chronic systemic steroids (more than 10mg prednisone or equivalent per day) or any form of immunosuppressive therapy within 7 days before the first administration of the study drug.

   Note: glucocorticoids are permitted for the following indications:
   * eye, intranasal or topical use.
   * inhalants for the management of asthma or chronic obstructive pulmonary disease.
   * systemic physiological corticosteroid replacement therapy for hormone replacement therapy, preventing vomiting, regulating symptoms suspected of immunological etiology, or as a pretreatment of IV contrast agent allergy or chemotherapeutic agent.

     16 Active autoimmune diseases requiring systemic treatment (i.e. use of disease regulating drugs, corticosteroids or immunosuppressants) in the past 2 years. Alternative treatment (e.g., thyroxine, insulin or physiological corticosteroid replacement treatment due to adrenal or pituitary insufficiency) is not considered systemic treatment and is allowed.

     17 Currently or previously participated in the study of investigational drugs, or used investigational devices within 4 weeks before the first administration of the study intervention. Note: subjects who have entered the follow-up period of the experimental study can participate in this study as long as they are > 4 weeks after the last administration of previous research drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-06-21 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 2 years
  Progression-free Survival is the time from the date of randomization until either documented disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China